CLINICAL TRIAL: NCT01892150
Title: Histologic Response to UVA and UVB Exposure During the Use of Sunscreen With Anti-inflammatory and Anti-oxidant Properties - A Pilot Study
Brief Title: Histologic Response to UVA and UVB Exposure During the Use of Sunscreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: Siriraj-Eucerin02; 721/2555(EC2) (Other: Siriraj Institutional Review Board)
Record Dates: First submitted 2013-05-23; First posted 2013-07-04 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Solar Elastosis
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunscreen (Experimental): Apply sunscreen before and after UVA and UVB irradiation
  Interventions: Other: Sunscreen

INTERVENTIONS:
Other: Sunscreen — Apply sunscreen before and after UVA and UVB irradiation

SUMMARY:
Anti-inflammatory and anti-oxidant agents have become the important ingredients in sunscreen. However, there is no histologic study about the effects of anti-inflammatory and anti-oxidative properties of sunscreen to prevent premature aging from UVA and UVB.

DETAILED DESCRIPTION:
Premature aging can be prevented by using sunscreen. Currently, anti-inflammatory and anti-oxidant agents have become the important ingredients in sunscreen. However, there is no histologic study about the effects of anti-inflammatory and anti-oxidative properties of sunscreen to prevent premature aging from UVA and UVB.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 35-65 years who were scheduled for abdominoplasty
* the excised area should be larger than 18x10 cm2
* no skin diseases or lesions on the excised area
* no topical treatment on excised area more than 1 month prior to this study

Exclusion Criteria:

* pregnancy
* lactation
* have tattoo or striae distensae on abdomen

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
H&E Staining | 2 Months
  Review difference in H&E staining in tissue biopsy before and after UVA / UVB irradiation

SECONDARY OUTCOMES:
Tyrosinase Staining | 2 Months
  Review difference in Tyrosinase staining in tissue biopsy before and after UVA / UVB irradiation to evaluate the effects of pigment darkening after UV exposure

OTHER OUTCOMES:
8-OH-dG Staining | 2 Months
  Review difference in 8-OH-dG staining in tissue biopsy before and after UVA / UVB irradiation to evaluate the quantity of free radical species after UV exposure
MMP1 Staining | 2 Months
  Review difference in MMP1 staining in tissue biopsy before and after UVA / UVB irradiation to evaluate the collagen and ground substances destruction after UV exposure

CONTACTS AND LOCATIONS:
Overall Officials: Rungsima Wanitphakdeedecha, MD, MA, MSc, Principal Investigator — Mahidol University
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Result] Lavker RM, Gerberick GF, Veres D, Irwin CJ, Kaidbey KH. Cumulative effects from repeated exposures to suberythemal doses of UVB and UVA in human skin. J Am Acad Dermatol. 1995 Jan;32(1):53-62. doi: 10.1016/0190-9622(95)90184-1. PMID 7822517